CLINICAL TRIAL: NCT01395134
Title: Randomized Controlled Trial of Visualization Versus Neuromonitoring of the External Branch of the Superior Laryngeal Nerve During Thyroidectomy.
Brief Title: Visualization Versus Neuromonitoring of the External Branch of the Superior Laryngeal Nerve During Thyroidectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jagiellonian University (Other)
Responsible Party: Piotr Laidler / Head of the Biomedical Research Committee of the Jagiellonian University, Biomedical Research Committee of the Jagiellonian University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BBN/501/ZKL/1446
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2011-07-15 (Estimated); Status verified 2011-07

CONDITIONS: Thyroid,; Goiter,
Keywords: External branch of the superior laryngeal nerve,; Recurrent laryngeal nerve,; Intraoperative neuromonitoring,; Thyroid surgery
MeSH Terms: conditions — Thyroid Diseases; Goiter

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Visualization of the EBSLN and RLN (No Intervention): Visual inspection of the nerves.
- Neuromonitoring of the EBSLN and RLN (Experimental): Electrical stimulation and monitoring of the nerves' function.
  Interventions: Device: Neuromonitoring

INTERVENTIONS:
Device: Neuromonitoring — Electrical stimulation of the nerve: 1 mA, 4 Hz with surface electromyography of the vocalis muscles.
  Other Names: IONM
  Arms: Neuromonitoring of the EBSLN and RLN

SUMMARY:
Injury to the external branch of the superior laryngeal nerve (EBSLN) during thyroidectomy results in lowered fundamental frequency of the voice and worsened voice performance in producing high-frequency sounds. It remains unclear if use of intraoperative nerve monitoring (IONM) can improve clinical outcome of thyroidectomy in terms of preserved individual voice performance. This study was designed to test that hypothesis.

DETAILED DESCRIPTION:
Phonation changes following thyroidectomy have been reported in many investigations. They are considered to be multifactorial in origin and can be a consequence of laryngeal nerve injury or other events during thyroidectomy including arytenoids trauma after endotracheal intubation, cricothyroid dysfunction, strap muscle malfunction or lesion of the perithyroidal neural plexus, laryngotracheal fixation with impairment of vertical movement and psychological reaction to the operation. Injury to the external branch of the superior laryngeal nerve (EBSLN) can occur during the dissection and clamping of the superior thyroid vessels and the prevalence of this complication has been reported from 0.5% to 58%. This injury causes a complete paralysis of the cricothyroid muscle which results in lowered fundamental frequency of the voice and worsened voice performance in producing high-frequency sounds. Intraoperative nerve monitoring (IONM) has gained widespread acceptance as an adjunct to the gold standard of visual nerve identification and this technique can be used to identify both the recurrent laryngeal nerve (RLN) and the EBSLN. However, it remains unclear if there is any IONM added-value to the clinical outcome of thyroidectomy in terms of preserved individual voice performance. This study was designed to test that hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* thyroid pathology qualified for first-time bilateral neck surgery in a female patient with small to moderate sized goiter (below 100 ml in volume).

Exclusion Criteria:

* male gender,
* previous neck surgery,
* unilateral thyroid pathology eligible for unilateral lobectomy,
* goiter volume above 100 ml,
* preoperatively diagnosed RLN palsy,
* abnormal preoperative voice assessment on GRBAS scale,
* pregnancy or lactation,
* age below 18 years,
* high-risk patients ASA 4 grade (American Society of Anesthesiology),
* inability to comply with the scheduled follow-up protocol.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The identification rate of the external branch of the superior laryngeal nerve. | up to 6 months postoperatively

SECONDARY OUTCOMES:
Anatomical variability of the external branch of the superior laryngeal nerve according to Cernea classification. | up to 6 months postoperatively
The changes in postoperative voice performance. | up to 6 months postoperatively
  The voice assessment included pre- and postoperative videostrobolaryngoscopy and analysis of maximum phonation time (MPT), voice level (VL), fundamental frequency (Fo), and voice quality rating on GRBAS scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Barczynski, MD, PhD, Principal Investigator — Jagiellonian University, College of Medicine
Locations (1):
- Jagiellonian University, College of Medicine, Department of Endocrine Surgery, 3rd Chair of General Surgery, Krakow, Poland

REFERENCES:
- [Background] Cernea CR, Ferraz AR, Furlani J, Monteiro S, Nishio S, Hojaij FC, Dutra Junior A, Marques LA, Pontes PA, Bevilacqua RG. Identification of the external branch of the superior laryngeal nerve during thyroidectomy. Am J Surg. 1992 Dec;164(6):634-9. doi: 10.1016/s0002-9610(05)80723-8. PMID 1463114
- [Background] Cernea CR, Ferraz AR, Nishio S, Dutra A Jr, Hojaij FC, dos Santos LR. Surgical anatomy of the external branch of the superior laryngeal nerve. Head Neck. 1992 Sep-Oct;14(5):380-3. doi: 10.1002/hed.2880140507. PMID 1399571
- [Background] Randolph GW, Dralle H; International Intraoperative Monitoring Study Group; Abdullah H, Barczynski M, Bellantone R, Brauckhoff M, Carnaille B, Cherenko S, Chiang FY, Dionigi G, Finck C, Hartl D, Kamani D, Lorenz K, Miccolli P, Mihai R, Miyauchi A, Orloff L, Perrier N, Poveda MD, Romanchishen A, Serpell J, Sitges-Serra A, Sloan T, Van Slycke S, Snyder S, Takami H, Volpi E, Woodson G. Electrophysiologic recurrent laryngeal nerve monitoring during thyroid and parathyroid surgery: international standards guideline statement. Laryngoscope. 2011 Jan;121 Suppl 1:S1-16. doi: 10.1002/lary.21119. PMID 21181860
- [Background] Lifante JC, McGill J, Murry T, Aviv JE, Inabnet WB 3rd. A prospective, randomized trial of nerve monitoring of the external branch of the superior laryngeal nerve during thyroidectomy under local/regional anesthesia and IV sedation. Surgery. 2009 Dec;146(6):1167-73. doi: 10.1016/j.surg.2009.09.023. PMID 19958945
- [Background] Bellantone R, Boscherini M, Lombardi CP, Bossola M, Rubino F, De Crea C, Alesina P, Traini E, Cozza T, D'alatri L. Is the identification of the external branch of the superior laryngeal nerve mandatory in thyroid operation? Results of a prospective randomized study. Surgery. 2001 Dec;130(6):1055-9. doi: 10.1067/msy.2001.118375. PMID 11742338
- [Derived] Barczynski M, Konturek A, Stopa M, Honowska A, Nowak W. Randomized controlled trial of visualization versus neuromonitoring of the external branch of the superior laryngeal nerve during thyroidectomy. World J Surg. 2012 Jun;36(6):1340-7. doi: 10.1007/s00268-012-1547-7. PMID 22402975